CLINICAL TRIAL: NCT04950621
Title: Comparison of Efficacy and Safety of Remimazolam and Propofol in Patients Undergoing Endovascular Procedures of Cerebrovascular Disorders: A Single-center,Randomized,Single-blind, Non-inferiority Trial
Brief Title: Remimazolam and Endovascular Procedures of Cerebrovascular Diseases
Acronym: REPEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-20201225
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cerebrovascular Disorders; Anesthesia
Keywords: propofol; Remimazolam; Endovascular Procedures
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization is done by an investigator who is not involved in anesthesia and outcome assessment. Participants are unaware of the group allocation. Due to the different color of remimazolam and propofol, the care provider is not blinded to the group allocation. At the end of the surgery, anesthetics are removed before outcome assessment. And the outcome assessor is blinded to the grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Experimental): In remimazolam group, a 0.1 mg/kg dose of intravenous remimazolam was administered for induction, and 0.3-0.7 mg/kg/h infusion for maintenance after intubation.
  Interventions: Drug: remimazolam
- Propofol (Active Comparator): In propofol group, a 2 mg/kg dose of intravenous propofol was administered for induction, and 4-12 mg/kg/h infusion for maintenance after intubation.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: remimazolam — Remimazolam will be administered during induction and maintenance for general anesthesia.
  Arms: Remimazolam
Drug: propofol — Propofol will be administered during induction and maintenance for general anesthesia.
  Arms: Propofol

SUMMARY:
Remimazolam, a novel ultra-short acting benzodiazepine that combined the advantages of midazolam and remifentanil, has been developed for procedural sedation, induction and maintenance of general anesthesia, and sedation in the ICU. Previous studies have suggested that efficacy and safety of remimazolam are not inferior to propofol or midazolam in patients undergoing colonoscopy,bronchoscopy and some other treatments. However, the efficacy and potential adverse effects of remimazolam on patients undergoing endovascular procedures of cerebrovascular disorders is still unclear. In this study, we tend to conduct a single-center, randomized, single-blind ,non-inferiority trial to compare the efficacy and safety of remimazolam and propofol in endovascular procedures of cerebrovascular disorders.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older
2. scheduled for interventional neurosurgery of cerebrovascular disorders under general anesthesia

Exclusion Criteria:

1. American Society of Anesthesiologists class Ⅲ or higher
2. Hunt-Hess class Ⅲ or higher
3. body mass index (BMI) < 18 kg/㎡ or > 30kg/㎡
4. large or giant cerebral aneurysms with diameters greater than 15mm and minor cerebral aneurysms with diameters less than 3mm
5. posterior circulation infarction
6. recurrence of an cerebral aneurysms after endovascular procedures or surgical clipping
7. severe abnormal coagulation function, severe liver and kidney function damage, or combined with heart and respiratory system failure
8. be allergic or likely to be allergic to the study drugs
9. participate in other clinical researchers within 3 months
10. history of neurological or psychiatric diseases
11. existed or suspected abuse of drug or alcohol
12. use of sedative or analgesics before surgery
13. patients with difficulty in communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
time to open eye | from the stop of trial drugs to open eye to verbal command, at an average of 15 minutes

SECONDARY OUTCOMES:
time to loss of consciousness | from initial administration of trial drugs to loss of response to verbal command, at an average of 5 minutes
time to recovery of spontaneous breathing | from end of giving trial drugs to recovery of spontaneous breathing ,at an average of 20 minutes
time to endotracheal tube extubation | from end of giving trial drugs to removing endotracheal tube ,at an average of 25 minutes
time to orientation | from end of giving trial drugs to recovery of orientation to name, location or date ,at an average of 30 minutes
the dosages of vasoactive drugs during surgery | from initial administration of trial drugs to end of surgery, at an average of 3 hours
Number of episodes of hypotension during surgery | from initial administration of trial drugs to end of surgery, at an average of 3 hours
  Hypotension is defined as decrease of mean arterial pressure more than 20% of the baseline, persisting longer than 1 minute
Number of episodes of hypertension during surgery | from initial administration of trial drugs to end of surgery, at an average of 3 hours
  Hypertension is defined as increase of mean arterial pressure more than 20% of the baseline, persisting longer than 1 minute
the level of lactic acid of arterial blood | at the end of the surgery
The highest Richmond Agitation and Sedation Score during emergence | from end of the surgery to 30 minutes after extubation, approximately 50 minutes
Renkin's Score at 30 days and three months after surgery | 30 days and three months after surgery
Glasgow outcome Score at discharge | at discharge, approximately 3 days after surgery
length of postoperative ICU stay and hospital stay | from entering the ICU to leaving the ICU and from admission to discharge, approximately 3 days
the incidence of major complications during postoperative hospitalization | from the end of surgery to discharge, approximately 3 days
the incidence of delirium during emergence | from end of surgery to 30 minutes after extubation
the incidence of delirium within 3 days after surgery | from end of surgery to 3 days after surgery
the level of serum interleukin-6, tumor necrosis factor-α and S100β | at the end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
individual data including protocol and statistical analysis plan will be shared during 3 months and 5 years following article publication after deidentification
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] Sneyd JR, Rigby-Jones AE. Remimazolam for anaesthesia or sedation. Curr Opin Anaesthesiol. 2020 Aug;33(4):506-511. doi: 10.1097/ACO.0000000000000877. PMID 32530890
- [Result] Keam SJ. Remimazolam: First Approval. Drugs. 2020 Apr;80(6):625-633. doi: 10.1007/s40265-020-01299-8. PMID 32274703
- [Result] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760